CLINICAL TRIAL: NCT01559051
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Intra-venous and Inhalation Implantation of Autologous Adipose-Derived Stromal Vascular Fraction Cells in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Safety and Efficacy of Adipose Derived Stem Cells for Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-COPD-001
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary; Lungs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Anesthesia, Local; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Injection and Inhalation infusion of AD-SVF (Experimental): AD-SVF harvested from Autologous Adipose Tissue will be deliver after processing via IV and Inhalation
  Interventions: Procedure: Lipoaspiration with Local anesthesia

INTERVENTIONS:
Procedure: Lipoaspiration with Local anesthesia — Patients undergo a liposuction under local Anethesia. The AD-SVF are then isolated and infused IV and by inhalation delivery.
  Other Names: Liposuction

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the health of patients with human Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of Autologous SVF (AD-SVF) implantation after liposuction using an IV delivery system and Inhalation infusion. AD-SVF will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered intravenously.

The adipose tissue specimen will be collected from the patient's abdomen or applicable area using tumescent syringe liposuction. The adipose tissue is transferred to the laboratory for separation of the adipose tissue-derived stem cells, which are then transferred for IV delivery. The number of cells injected will vary depending on the amount of tissue processed and the number of cells obtained from the process.

ELIGIBILITY:
Inclusion Criteria:

* A prior diagnosis of moderate or severe COPD
* GOLD III and IV
* Age between 25 and 80 years
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. will have an expert consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Severe asthma that would contraindicate surgery
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity improved compared to baseline | 3 months, 6 months
  6 Minute Walk Test
Number of adverse events | 3 months, 6 months

SECONDARY OUTCOMES:
Quality of Life improved compared to baseline | 3 months, 6 months
  St. George Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided